CLINICAL TRIAL: NCT01358266
Title: A Phase III, Multinational, Multicenter, Randomized, Double-Masked, Study for the Treatment of Active, Non-Infectious Uveitis of the Posterior Segment of the Eye
Brief Title: Study Assessing Double-masked Uveitis Treatment
Acronym: SAKURA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 32-007
Record Dates: First submitted 2011-05-19; First posted 2011-05-23 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-06

CONDITIONS: Uveitis; Posterior, Disorder
MeSH Terms: conditions — Uveitis | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ophthalmic solution low dose (Active Comparator)
  Interventions: Drug: DE-109 44 ug
- Ophthalmic solution medium dose (Active Comparator)
  Interventions: Drug: DE-109 440 ug
- Ophthalmic solution high dose (Active Comparator)
  Interventions: Drug: DE-109 880 ug

INTERVENTIONS:
Drug: DE-109 44 ug — Low dose
  Other Names: Sirolimus
  Arms: Ophthalmic solution low dose
Drug: DE-109 440 ug — Medium dose
  Other Names: Sirolimus
  Arms: Ophthalmic solution medium dose
Drug: DE-109 880 ug — High dose
  Other Names: Sirolimus
  Arms: Ophthalmic solution high dose

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of intravitreal injections of DE-109 ophthalmic solution.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of active uveitis
* 18 years of age or older
* Sign informed consent
* Meet best corrected ETDRS visual acuity

Exclusion Criteria:

* Uveitis of infectious etiology
* Suspected/confirmed central nervous system or ocular lymphoma
* Primary diagnosis of anterior uveitis
* Uncontrolled glaucoma
* Use of topical oculary medication
* Implanted device
* Significant ocular disease
* Lens/media opacities or obscured ocular media
* Intraocular surgery or treatments
* Capsulotomy
* Ocular or periocular infection
* Pupillary dilation
* History of herpetic infection
* Toxoplasmosis or toxoplasmosis scar
* Ocular malignancy
* Allergy or hypersensitivity to study drug
* Participation in other uveitis trial within 30 days
* Monoclonal antibody treatment or biologic therapy
* Any systemic condition/infection
* Immunosuppressive therapy or immunocompromised
* Malignancy remission
* Females who are pregnant or lactating and females not using adequate contraceptives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2011-05; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abu Abraham, MD, Study Director — Santen Inc.
Locations (151):
- United States (74):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Beverly Hills, California
  - Loma Linda, California
  - Los Angeles, California
  - Mountain View, California
  - Sacramento, California
  - Torrance, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Golden, Colorado
  - Altamonte Springs, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Winter Haven, Florida
  - Augusta, Georgia
  - Chicago, Illinois
  - Oak Park, Illinois
  - Indianapolis, Indiana
  - Iowa City, Iowa
  - Wichita, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Peabody, Massachusetts
  - Ann Arbor, Michigan
  - Grand Rapids, Michigan
  - Jackson, Michigan
  - Royal Oak, Michigan
  - Southfield, Michigan
  - Edina, Minnesota
  - St Louis, Missouri
  - Missoula, Montana
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Portsmouth, New Hampshire
  - New Brunswick, New Jersey
  - Newark, New Jersey
  - Northfield, New Jersey
  - Teaneck, New Jersey
  - Toms River, New Jersey
  - Albany, New York
  - New York, New York
  - Orchard Park, New York
  - Rochester, New York
  - Slingerlands, New York
  - Southern Pines, North Carolina
  - Winston-Salem, North Carolina
  - Cleveland, Ohio
  - Eugene, Oregon
  - Camp Hill, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Reading, Pennsylvania
  - West Mifflin, Pennsylvania
  - Columbia, South Carolina
  - Ladson, South Carolina
  - Rapid City, South Dakota
  - Knoxville, Tennessee
  - Arlington, Texas
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Richmond, Virginia
  - Virginia Beach, Virginia
  - Milwaukee, Wisconsin
- Argentina (6):
  - Buenos Aires
  - Mendoza
  - Olivos
  - Pilar
  - Rosario
  - San Juan Bautista
- Austria (2):
  - Graz
  - Klagenfurt
- Brazil (7):
  - Americana
  - Araraquara
  - Londrina
  - Recife
  - Rio de Janeiro
  - São Paulo
  - Sorocaba
- Santiago, Chile
- Colombia (4):
  - Bogotá
  - Cali
  - Floridablanca
  - Medellín
- France (3):
  - Marseille
  - Nantes
  - Paris
- Germany (7):
  - Berlin
  - Cologne
  - Freiburg im Breisgau
  - Heidelberg
  - München
  - Münster
  - Tübingen
- India (10):
  - Ahmedabad
  - Bangalore
  - Bhubaneshwar
  - Chennai
  - Hyderabad
  - Kolkata
  - Madurai
  - Mumbai
  - New Delhi
  - Noida
- Israel (8):
  - Afula
  - Beersheba
  - Haifa
  - Jerusalem
  - Petah Tikva
  - Ramat Gan
  - Rehovot
  - Tel Aviv
- Italy (6):
  - Bologna
  - Florence
  - Milan
  - Padua
  - Pisa
  - Reggio Emilia
- Japan (5):
  - Hokkaido
  - Osaka
  - Sapporo
  - Sendai
  - Tokyo
- Peru (2):
  - Lima
  - Trujillo
- Poland (4):
  - Lodz
  - Lublin
  - Poznan
  - Wroclaw
- Spain (5):
  - Alicante
  - Barcelona
  - Madrid
  - Santiago de Compostela
  - Torrevieja
- Turkey (Türkiye) (3):
  - Ankara
  - Istanbul
  - Izmir
- United Kingdom (4):
  - Belfast
  - Bradford
  - Bristol
  - London

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects who entered open-label period are defined as subjects who received at least one open-label injection during the open-label treatment period (Month 6 to Month 12, exclude Amendment 2 subjects), or those who had entered the open-label retreatment period (Month 12 to Month 24) with or without any PRN injections.
Groups:
- DE-109 44 μg; DE-109 440 μg: SAKURA Study 1 & Study 2 (Amendment #2) Double-Masked Treatment Period Injection on Day 1, Month 2, Month 4 Double-Masked PRN Treatment Period May receive up to 3 injections PRN from Month 6 through Month 10 SAKURA Study 1 & Study 2 (Amendments #3 and #4) Injection on Day 1, Month 2, Month 4 SAKURA Study 2 (Amendment #5) Double-Masked Treatment Period Injection on Day 1, Month 2, Month 4
- DE-109 880 μg: SAKURA Study 1 & Study 2 (Amendment #2) Double-Masked Treatment Period Injection on Day 1, Month 2, Month 4 Double-Masked PRN Treatment Period May receive up to 3 injections PRN from Month 6 through Month 10 SAKURA Study 1 & Study 2 (Amendments #3 and #4) Injection on Day 1, Month 2, Month 4
  Open-Label Treatment Period Injection on Month 6, Month 8, Month 10 Open-Label Re-Treatment Period May receive up to 6 injections PRN through Month 22 SAKURA Study 2 (Amendment #5) Double-Masked Treatment Period Injection on Day 1, Month 2, Month 4
Period: Double-Masked Period
Arm/Group | DE-109 44 μg | DE-109 440 μg | DE-109 880 μg
Started | 208 | 208 | 176
Completed | 175 | 162 | 137
Not Completed | 33 | 46 | 39
Period: Open-Label Period
Arm/Group | DE-109 44 μg | DE-109 440 μg | DE-109 880 μg
Started | 119 | 102 | 114
Completed | 63 | 58 | 44
Not Completed | 56 | 44 | 70

BASELINE CHARACTERISTICS:
Groups:
- DE-109 44 µg: Double Masked Phase Low Dose 44 µg Open Label Phase High Dose 880 µg
- DE-109 440 µg: Double Masked Phase Medium Dose 440 µg Open Label Phase High Dose 880 µg
- DE-109 880 µg: Double Masked Phase High Dose 880 µg Open Label Phase High Dose 880 µg
- Total: Total of all reporting groups
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg | Total
Number analyzed (Participants) | 208 | 208 | 176 | 592
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 188 | 191 | 153 | 532
  >=65 years | 20 | 17 | 23 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 117 | 113 | 343
  Male | 95 | 91 | 63 | 249
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 1 | 3 | 8
  Asian | 76 | 77 | 72 | 225
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 0 | 2
  Black or African American | 16 | 13 | 13 | 42
  White | 93 | 99 | 79 | 271
  More than one race | 8 | 7 | 3 | 18
  Unknown or Not Reported | 10 | 10 | 6 | 26
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 4 | 4 | 5 | 13
  Argentina | 20 | 13 | 10 | 43
  United States | 70 | 71 | 45 | 186
  Japan | 4 | 8 | 6 | 18
  United Kingdom | 4 | 8 | 4 | 16
  India | 69 | 65 | 65 | 199
  Spain | 0 | 1 | 2 | 3
  Austria | 3 | 2 | 0 | 5
  Turkey | 4 | 2 | 0 | 6
  Brazil | 2 | 3 | 5 | 10
  Poland | 1 | 3 | 2 | 6
  Italy | 2 | 7 | 2 | 11
  Israel | 7 | 1 | 3 | 11
  Chile | 3 | 2 | 4 | 9
  France | 4 | 3 | 7 | 14
  Peru | 6 | 10 | 10 | 26
  Germany | 5 | 5 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint, VH 0 Response, Was Defined as Having a VH Score of 0 at Month 5
Description: At each visit, slit-lamp biomicroscopy was used to assess VH and opacification. For slit-lamp biomicroscopy, a contact or non-contact lens could have been used. The modified SUN scale for VH was used to measure VH and opacification
  Vitreous Haze Scale Description VH score 0 = No inflammation
Time Frame: Day1 (Baseline) and Month 5 (Day150)
Measure: Count of Participants; unit: Participants
Groups:
- DE-109 44 µg: Low Dose DE-109 44 µg
- DE-109 440 µg: Medium Dose DE-109 440 µg
- DE-109 880 µg: High Dose DE-109 880 µg
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg
Number analyzed (Participants) | 208 | 208 | 176
Participants | 28 | 44 | 27

2. Secondary Outcome: VH 0 or 2-unit Response: Having a Reduction (Improvement) of at Least 2 Units From Baseline in VH Score or a VH Score of 0 at Month 5 (Modified SUN Scale)
Description: At each visit, slit-lamp biomicroscopy was used to assess VH and opacification. For slit-lamp biomicroscopy, a contact or non-contact lens could have been used. The modified SUN scale for VH was used to measure VH and opacification Vitreous Haze Scale Step Description 0 No inflammation 0.5+ Trace Inflammation (slight blurring of the optic disc margins and or loss of nerve fiber layer reflex)
  1. Mild blurring of the retinal vessels and optic nerve 1.5+ Optic nerve head and posterior retina view obstruction greater than 1+ but less than 2+
  2. Moderate blurring of the optic nerve head
  3. Marked blurring of the optic nerve head
  4. Optic Nerve head not visible
Time Frame: Day1/Baseline and Day150/Month 5
Measure: Count of Participants; unit: Participants
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg
Number analyzed (Participants) | 208 | 208 | 176
Participants | 43 | 56 | 33

3. Secondary Outcome: VH 0 or 0.5+ Response: Having a VH Score of 0 or 0.5+ at Month 5 (Modified SUN Scale)
Description: At each visit, slit-lamp biomicroscopy was used to assess VH and opacification. For slit-lamp biomicroscopy, a contact or non-contact lens could have been used. The modified SUN scale for VH was used to measure VH and opacification Vitreous Haze Scale Description VH score 0.5+=Trace Inflammation (slight blurring of the optic disc margins and or loss of nerve fiber layer reflex)
Time Frame: Day1/Baseline and Day150/Month 5
Measure: Count of Participants; unit: Participants
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg
Number analyzed (Participants) | 208 | 208 | 176
Participants | 84 | 104 | 70

4. Other Pre Specified Outcome: VH 0 Response at Month 6: Having a VH Score of 0 at Month 6 (Modified SUN Scale)
Description: as for outcome 1
Time Frame: Day1/Baseline and Day180/Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg
Number analyzed (Participants) | 208 | 208 | 176
Participants | 29 | 43 | 51

5. Other Pre Specified Outcome: VH 0 or 2-unit Response at Month 6: Having a VH Score of 0 or a Decrease (Improvement) of at Least 2 Units From Baseline in VH Score at Month 6 (Modified SUN Scale)
Description: as for outcome 2
Time Frame: Day1/Baseline and Day180/Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg
Number analyzed (Participants) | 208 | 208 | 176
Participants | 42 | 52 | 26

6. Other Pre Specified Outcome: VH 0 or 0.5+ Response at Month 6: Having a VH Score of 0 or 0.5+ at Month 6 (Modified SUNscale)
Description: as for outcome 2
Time Frame: Day1/Baseline and Day180/Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | DE-109 44 µg | DE-109 440 µg | DE-109 880 µg
Number analyzed (Participants) | 208 | 208 | 176
Participants | 81 | 90 | 66

ADVERSE EVENTS:
Time Frame: Adverse events - begin capturing once the first treatment is given. Per Schedule of Events through study completion, up to 24 months.
Description: Any subject with multiple AEs of one system organ class is counted only once for that class.
  Subjects are classified by actual treatment received. AEs summaries were done with the Safety Population (N=590) defined as all randomized subjects who received at least one study treatment.1 subject was randomized to the 44 μg dose group but received 880 μg at Month 2
  1subject was randomized to the 44 μg dose group but received 880 μg at Month 4 both subjects are reflected in the 880/880 μg group.
Groups:
- DE-109 44 µg - Double Masked: Double Masked Phase Low Dose 44 µg
- DE-109 440 µg - Double Masked: Double Masked Phase Medium Dose 440 µg
- DE-109 880 µg - Double Masked: Double Masked Phase High Dose 880 µg
- DE-109 880 µg - Open-Label: Open-label Phase High Dose 880 µg
Arm/Group | DE-109 44 µg - Double Masked | DE-109 440 µg - Double Masked | DE-109 880 µg - Double Masked | DE-109 880 µg - Open-Label
All-Cause Mortality (participants affected / at risk) | 1/207 | 0/205 | 0/178 | 0/321
Serious Adverse Events (participants affected / at risk) | 41/207 | 45/205 | 38/178 | 59/321
Other Adverse Events (participants affected / at risk) | 165/207 | 166/205 | 148/178 | 210/321
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DE-109 44 µg - Double Masked (N=207) | DE-109 440 µg - Double Masked (N=205) | DE-109 880 µg - Double Masked (N=178) | DE-109 880 µg - Open-Label (N=321)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — 1 subject 44 µg dose group died • a 63-year-old male who suffered a stroke on Day 54 (11 Sep 2012) of study participation.This subject died on Study Day 55 (12 Sep 2012). This SAE was reported as severe, and not related to the study medication.
Uveitis (Eye disorders) | 6 (7) | 10 (12) | 13 (13) | 5 (7)
Choroiditis (Eye disorders) | 8 (8) | 4 (4) | 3 (4) | 6 (7)
Cataract (Eye disorders) | 4 (4) | 2 (2) | 3 (4) | 4 (6)
Non-infectious endophthalmitis (Eye disorders) | 0 (0) | 1 (1) | 7 (7) | 11 (11)
Iridocyclitis (Eye disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0)
Retinal detachment (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Visual acuity reduced (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Vitritis (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 4 (4)
Cystoid macular oedema (Eye disorders) | 2 (2) | 1 (2) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Intermediate uveitis (Eye disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Macular oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Optic atrophy (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Anterior chamber inflammation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal deposits (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal epithelium defect (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Corneal oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye haemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ocular vasculitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Open angle glaucoma (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal infiltrates (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal oedema (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Eye infection toxoplasmal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratitis herpetic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure increased (Investigations) | 3 (3) | 3 (3) | 3 (3) | 3 (3)
Fibrin (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraocular pressure decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medication residue (General disorders) | 2 (2) | 2 (2) | 4 (5) | 6 (10)
Device dislocation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Central nervous system lymphoma (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Glaucoma (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Optic Neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DE-109 44 µg - Double Masked (N=207) | DE-109 440 µg - Double Masked (N=205) | DE-109 880 µg - Double Masked (N=178) | DE-109 880 µg - Open-Label (N=321)
Iridocyclitis (Eye disorders) | 31 (41) | 32 (46) | 30 (51) | 31 (48)
Uveitis (Eye disorders) | 19 (23) | 15 (18) | 29 (42) | 15 (16)
Conjunctival haemorrhage (Eye disorders) | 22 (32) | 19 (22) | 26 (33) | 24 (33)
Eye pain (Eye disorders) | 18 (20) | 22 (27) | 19 (22) | 14 (17)
Intermediate uveitis (Eye disorders) | 16 (21) | 15 (21) | 14 (20) | 9 (14)
Cataract (Eye disorders) | 11 (13) | 8 (9) | 13 (13) | 32 (33)
Cystoid macular oedema (Eye disorders) | 12 (18) | 15 (17) | 11 (12) | 7 (7)
Choroiditis (Eye disorders) | 11 (14) | 11 (15) | 5 (6) | 6 (8)
Cataract subcapsular (Eye disorders) | 3 (3) | 10 (10) | 12 (13) | 17 (18)
Macular oedema (Eye disorders) | 3 (3) | 11 (14) | 9 (11) | 8 (8)
Intraocular pressure increased (Investigations) | 34 (50) | 34 (62) | 43 (64) | 44 (62)
Headache (Nervous system disorders) | 7 (9) | 12 (14) | 4 (4) | 7 (8)
Conjunctival hyperaemia (Eye disorders) | 11 (13) | 11 (12) | 6 (9) | 13 (14)
Vitreous opacities (Eye disorders) | 5 (5) | 5 (8) | 9 (13) | 9 (12)
Dry eye (Eye disorders) | 12 (13) | 4 (4) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No